CLINICAL TRIAL: NCT03537534
Title: Intraurethral Lidocaine After Endourology Procedure to Improve Dysuria in Anesthetized Patients
Brief Title: Intraurethral Lidocaine After Endourology Procedures
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: San Antonio Uniformed Services Health Education Consortium (U.S. Federal Agency)
Responsible Party: Principal Investigator, Christopher Allam, Director of Endourology and Laparoscopy, San Antonio Uniformed Services Health Education Consortium
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: C.2018.055d
Record Dates: First submitted 2018-05-15; First posted 2018-05-25 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Dysuria
MeSH Terms: conditions — Dysuria | interventions — phenylmercury borate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Experiment (Experimental): Lidocaine jelly (2%) 5mL x 1 dose only
  Interventions: Drug: Lidocaine Jet Injector
- Placebo (Placebo Comparator): Surgilube 5mL x 1 dose only
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Lidocaine Jet Injector — Applying Lidocaine following endourologic procedure
  Other Names: Urojet
  Arms: Experiment
Drug: Placebos — Applying surgilube following endourologic procedure
  Other Names: Surgilube
  Arms: Placebo

SUMMARY:
Many urological conditions are diagnosed and treated with the use of endourology procedures. Unfortunately, dysuria is a common patient complaint following these procedures. Intraurethral lidocaine instillation is regularly used prior to office-based endourology procedures to alleviate dysuria, as well as, discomfort during the procedure.. Studies have confirmed that office-based procedures using intraurethral lidocaine have resulted in less patient reported dysuria. Many endourology procedures are done under general anesthesia such as urinary stone treatments or resection of bladder tumors. There is a paucity of data regarding the use of intraurethral lidocaine at the conclusion of these procedures evaluating patient reported dysuria. We have designed a prospective, randomized, placebo controlled trial to evaluate the role of intraurethral lidocaine instillation following endourology procedures in the anesthetized patient.

ELIGIBILITY:
Inclusion Criteria: Adult patients, age 18 and older scheduled to undergo endourologic procedure to include ureteroscopy, rigid diagnostic cystoscopy, bladder biopsy, laser lithotripsy, cystolithalopaxy, and transurethral resection of bladder tumor in the operating room under general anesthesia.

-

Exclusion Criteria: active urinary tract infection, current dysuria symptoms, pregnant females, urethral stricture disease, indwelling foley catheter, and history of pelvic radiation

-

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-04-15 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Subjective patient symptom score | 1 day (immediately before and after procedure)
  questionnaire scores

SECONDARY OUTCOMES:
Patient complications | within 30 days
  Unplanned patient returns to clinic or ED, UTIs, admissions

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Allam, DO, Principal Investigator — San Antonio Uniformed Services Health Education Consortium
Locations (1):
- BAMC, Fort Sam Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No